CLINICAL TRIAL: NCT05449379
Title: Evaluation of Influence of Proprietary Physical Training Program on Quality of Life, Physical Endurance, Function of Muscles and Myokines Profile in Patients After COVID-19 Infection.
Brief Title: Evaluation of Effectiveness of Proprietary Rehabilitation Program in Patients After COVID-19 Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SUB/1/DN/22/001/3309
Record Dates: First submitted 2022-07-07; First posted 2022-07-08 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; Rehabilitation
Keywords: COVID-19; rehabilitation; respiratory training
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be double blind, patients will be unaware of being assigned to a group and investigators assessing functional state in the next stages of the study will not conduct rehabilitation and will not be aware of the allocation of patients to groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post COVID experimental group (Experimental): Safe protocol of 6 week physical training (aerobic training, resistance training, general improvement training, stretching training and respiratory rehabilitation) adjusted to the clinical state of patients plus additional resistance respiratory training with the use of respiratory muscle trainer (Philips Respironics Threshold IMT).
  Interventions: Other: Respiratory training with the use of resistance set on respiratory muscle trainer
- Post COVID control group (Placebo Comparator): Safe protocol of 6 week physical training (aerobic training, resistance training, general improvement training, stretching training and respiratory rehabilitation) adjusted to the clinical state of patients. No resistance set on respiratory muscle trainer (Philips Respironics Threshold IMT).
  Interventions: Other: Respiratory training without resistance set on respiratory muscle trainer

INTERVENTIONS:
Other: Respiratory training with the use of resistance set on respiratory muscle trainer — Performing respiratory training with resistance set on respiratory trainer.
  Arms: Post COVID experimental group
Other: Respiratory training without resistance set on respiratory muscle trainer — Performing respiratory training with no resistance set on respiratory trainer
  Arms: Post COVID control group

SUMMARY:
The aim of the study is to evaluate the influence of 6 week physical training and respiratory rehabilitation performed in outpatients rehabilitation clinic on quality of life, symptoms, physical endurance, mental state, force of respiratory and skeletal muscles and myokines profile in patients after COVID-19 infection.

DETAILED DESCRIPTION:
The study of interventional, prospective character will be conducted in Rehabilitation Department of Medical University of Bialystok on total group of 60 participants less than 12 months after COVID-19 (coronavirus disease) infection. In all participants medical anamnesis, physical examination (including chest wall mobility), anthropometric measures, The Short Physical Performance Battery (SPPB), 6-minute walking test (6MWT six minute walking test) and treadmill stress test will be performed.

Medical history will consist of questions regarding course of COVID-19 and its consequences with special emphasis on dyspnea during daily activities in Borg scale and dyspnea in daily living in mMRC scale, coexisting diseases, treatment, lifestyle, etc. Quality of life will be assessed with use of The Short Form (36) Health Survey - SF-36), Post-COVID-19 Functional Status (PCFS] scale and Modified Fatigue Impact Scale (MFIS). Mental status will be evaluated with the use of Beck Depression Inventory (BDI) and Hamilton Depression Scale (HAMD)) Biochemical measures will be performed including, among others, myokines such as BDNF (brain-derived neurotrophic factor), adiponectin, fibroblast growth factor 21 (FGF21), resistin, myonectin and inflammatory markers, such as interleukin 6 ((Il-6), C-reactive protein (CRP).

Fasting venous blood will be collected in 2 tubes each a 10 ml, one dedicated to obtain serum ("on clot"), second with heparin) to perform biochemical analyses, In clinical evaluation measurement of respiratory (inspiratory and expiratory) muscles force with use of device MicroRPM (respiratory pressure meter), hand grip strength with use of hand dynamometer (Jamar) and strength of quadriceps muscles with use of digital dynamometer (AXIS) will be performed. During first visit also ECG (electrocardiogram), six minute walking test and treadmill stress test will be done. All patients will have diaphragm ultrasound with measurement of diaphragm thickness.

Patient will be randomized to the control and interventional groups. Control group will be subjected to the safe protocol of 6 week physical training (aerobic training, resistance training, general improvement training, stretching training and respiratory rehabilitation) adjusted to the clinical state of patients. Additionally patients will be recommended to perform a set of exercises at home under a supervision of physiotherapist.

Patients from interventional group in addition to the training protocol will be subjected to additional resistance respiratory training with the use of respiratory muscle trainer (Philips Respironics Threshold IMT). Control group will have placebo with no resistance set on respiratory muscle trainer (Philips Respironics Threshold IMT). The study will be double blind, patients will be unaware of being assigned to a group and investigators assessing functional state in the next stages of the study will not conduct rehabilitation and will not be aware of the allocation of patients to groups. Physiotherapists conducting rehabilitation will receive detailed, individual guidelines regarding the training parameters of each patient. In addition, both groups will be educated on rules of safe physical activity and how to deal with troublesome symptoms.

Physical endurance (6 MWT, treadmill stress test), respiratory function, respiratory and peripheral muscle strength, other functional tests (SPPB), biochemical determinations, dyspnea (mMRC, Borg scale), quality of life (SF-36, PCFS, MFIS) mental state (BDI, HAMD), chest wall mobility and diaphragm ultrasound will be assessed at the beginning and end of the intervention. In addition, an analysis of the potential change in lifestyle of all patients will be carried out using accelerometry counting daily number of steps and assessing physical activity. Each patient will be equipped with basic exercise equipment and the necessary monitors of physical activity and vital signs to carry out the recommended activities at home (except for training units in the outpatient clinic). A reassessment of the long-term effects will be performed six months after the end of the exercises and will include 6 MWT, treadmill stress test, SPPB, spirometry, measurement of respiratory muscles force, handgrip strength, strength of quadriceps muscles, SF-36, PCFS, MFIS, BDI, HAMD, assessment of dyspnea in Borg scale during daily activities, mMRC, blood samples for biochemical analyses, ), chest wall mobility and diaphragm ultrasound . Patients in both groups will be monitored with the use of accelerometers in order to asses daily activity, daily number of steps within 7 days prior to intervention, after intervention and after observation period.

ELIGIBILITY:
Inclusion Criteria:

* COVID 19 infection confirmed with a positive PCR (polymerase chain reaction) SARS-CoV-2 (Severe Scute Respiratory Syndrome coronavirus type 2) test less than 12 moths prior to intervention
* more than 14 days from the day of obtaining a positive PCR test result for SARS-CoV-2 or discharge from hospital.
* mMRC (modified Medical Research Council) score ≥1
* age >18 years
* informed consent signed by patient to conduct the study

Exclusion Criteria:

* severe pulmonary disease (e.g. COPD)
* the functional state that makes it impossible to carry out the pre-examination and improvement program
* severe chest pain
* worsening dyspnea
* hemoptysis
* worsening dry cough
* syncope
* worsening oedema of extremities
* myocarditis (less than 6 months from acute phase)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical endurance improvement assessment of 6 MWT distance and outcome of treadmill stress test. | 6 months
  6-min walk test (6 MWT) is a exercise test that entails measurement of distance walked over a span of 6 minutes by patient good outcome > 500 m, bad outcome < 200 m.
  Treadmill stress test is performed with use of Bruce or ModBruce (modified Bruce) protocol, the outcome is measured in metabolic equivalents (METs) adjusted to the sex and age
Evaluation of quality of life | 6 months
  Quality of life measurement with SF36 (The Short Form (36) Health Survey, which is a 36-item, patient-reported survey of patient health.The Optum™ SF-36v2® Health Survey asks 36 questions to measure functional health and wellbeing from the patient's point of view. It is a practical, reliable and valid measure of physical and mental health that can be completed in five to ten minutes. The more number of points witness of better quality of life. Scores are calibrated so that 50 is the average score or norm. This norm-based score allows comparison among the three surveys and across the more than 19,000 studies published in the past 20 years. This bibliography includes studies of hundreds of diseases, conditions and populations, and greatly enhances the ability to interpret SF health survey data in new studies.Range 0-180 points
Force of respiratory muscles | 6 months
  Measurement of maximal inspiratory and expiratory pressure

SECONDARY OUTCOMES:
Spirometry | 6 months
  Measurement of basic parameters as VC (vital capacity), FEV1 (forced expiratory volume in 1 second), FEV1/VC (forced expiratory volume in 1 second//vital capacity) ratio
Force of quadriceps muscles | 6 months
  Measurement the force of quadriceps muscles
Handgrip strength | 6 months
  Measurement of handgrip strength
The Short Physical Performance Battery (SPPB) | 6 months
  Series of tests used to evaluate lower extremity function and mobility including the gait speed, chair stand and balance tests. Range 0-12 points, 0-6 low performance, 10-12 high performance;
Weight | 6 months
  measurement of weight in kilograms
Beck Depression Inventory (BDI) | 6 months
  21-item, self-report rating inventory measuring characteristic attitudes and symptoms of depression. (Range 0-63 ponts, 0-11 points no depression, 50-63 points- severe depression)
Hamilton Depression Scale (HAMD)) | 6 months
  Multiple-item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. (Range 0-50 ponts, 0-6points no depression, 25-50 points- severe depression)
Post-COVID-19 Functional Status [PCFS] scale. Range 0-4 0- no limitation of daily functioning, 4 severe limitation of daily functioning | 6 months
  Simple and rapid self-report scale allowing monitoring of the functional impact of the disease
Modified Fatigue Impact Scale (MFIS). | 6 months
  21-item scale measuring the impact of fatigue on a patient's daily life.Range 0-84 points. 0- no impact, 84 very severe impact
Modified Medical Research Council (mMRC) | 6 months
  Modified Medical Research Council (mMRC) most commonly used validated scale to assess dyspnea in daily living in chronic pulmonary diseases. Range 0-4, 0 grade dyspnea only with strenuous exercise, 4 patient too dyspneic to leave house or breathless when dressing
Chest wall mobility | 6 months
  Measurement of chest wall mobility at the level of the xiphoid process and the tenth rib
Diaphragm ultrasound | 6 months
  Measurement of diaphragm thickness in ultrasonography
Modified Borg scale | 6 months
  10 item scale describing dyspnea during daily activities (0- no dyspnea, 10 ver very severe dyspnea)
Concentration of CRP | 6 months
  Measurement of serum concentrations of CRP (C-reactive protein) mg/dl
Concentration of Il-6 | 6 months
  Measurement of serum concentrations of interleukin 6 (IL-6) pg/ml
Concentration of BDNF( brain-derived neurotrophic factor) | 6 months
  Measurement of serum concentrations of BDNF ng/ml
Concentration of adiponectin | 6 months
  Measurement of serum concentrations adiponectin ug/ml
Concentration of fibroblast growth factor 21 (FGF21) | 6 months
  Measurement of serum concentrations of fibroblast growth factor 21 (FGF21) ng/ml
Concentration of resistin | 6 months
  Measurement of serum concentrations resistin ng/ml
Concentration of myonectin | 6 months
  Measurement of serum concentrations myonectin ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kuryliszyn-Moskal, Professor, Study Chair — Medical University of Bialystok
Locations (1):
- Medical University of Bialystok, Department of Rehabilitation, Bialystok, Podlaskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu K, Zhang W, Yang Y, Zhang J, Li Y, Chen Y. Respiratory rehabilitation in elderly patients with COVID-19: A randomized controlled study. Complement Ther Clin Pract. 2020 May;39:101166. doi: 10.1016/j.ctcp.2020.101166. Epub 2020 Apr 1. PMID 32379637
- [Background] Dun Y, Liu C, Ripley-Gonzalez JW, Liu P, Zhou N, Gong X, You B, Du Y, Liu J, Li B, Liu S. Six-month outcomes and effect of pulmonary rehabilitation among patients hospitalized with COVID-19: a retrospective cohort study. Ann Med. 2021 Dec;53(1):2099-2109. doi: 10.1080/07853890.2021.2001043. PMID 34766857
- [Background] Benzarti W, Toulgui E, Prefaut C, Chamari K, Ben Saad H. General practitioners should provide the cardiorespiratory rehabilitation' 'minimum advice' for long COVID-19 patients. Libyan J Med. 2022 Dec;17(1):2009101. doi: 10.1080/19932820.2021.2009101. No abstract available. PMID 34839808
- [Background] Yan H, Ouyang Y, Wang L, Luo X, Zhan Q. Effect of respiratory rehabilitation training on elderly patients with COVID-19: A protocol for systematic review and meta-analysis. Medicine (Baltimore). 2020 Sep 11;99(37):e22109. doi: 10.1097/MD.0000000000022109. PMID 32925755
- [Background] Wang TJ, Chau B, Lui M, Lam GT, Lin N, Humbert S. Physical Medicine and Rehabilitation and Pulmonary Rehabilitation for COVID-19. Am J Phys Med Rehabil. 2020 Sep;99(9):769-774. doi: 10.1097/PHM.0000000000001505. PMID 32541352
- [Background] Spruit MA, Holland AE, Singh SJ, Tonia T, Wilson KC, Troosters T. COVID-19: interim guidance on rehabilitation in the hospital and post-hospital phase from a European Respiratory Society- and American Thoracic Society-coordinated international task force. Eur Respir J. 2020 Dec 3;56(6):2002197. doi: 10.1183/13993003.02197-2020. Print 2020 Dec. PMID 32817258
- [Background] Cheng YY, Chen CM, Huang WC, Chiang SL, Hsieh PC, Lin KL, Chen YJ, Fu TC, Huang SC, Chen SY, Chen CH, Chen SM, Chen HS, Chou LW, Chou CL, Li MH, Tsai SW, Wang LY, Wang YL, Chou W. Rehabilitation programs for patients with COronaVIrus Disease 2019: consensus statements of Taiwan Academy of Cardiovascular and Pulmonary Rehabilitation. J Formos Med Assoc. 2021 Jan;120(1 Pt 1):83-92. doi: 10.1016/j.jfma.2020.08.015. Epub 2020 Aug 17. PMID 32863084
- [Background] Azoulay D, Shehadeh M, Chepa S, Shaoul E, Baroum M, Horowitz NA, Kaykov E. Recovery from SARS-CoV-2 infection is associated with serum BDNF restoration. J Infect. 2020 Sep;81(3):e79-e81. doi: 10.1016/j.jinf.2020.06.038. Epub 2020 Jun 20. No abstract available. PMID 32569603
- [Background] Ajaz S, McPhail MJ, Singh KK, Mujib S, Trovato FM, Napoli S, Agarwal K. Mitochondrial metabolic manipulation by SARS-CoV-2 in peripheral blood mononuclear cells of patients with COVID-19. Am J Physiol Cell Physiol. 2021 Jan 1;320(1):C57-C65. doi: 10.1152/ajpcell.00426.2020. Epub 2020 Nov 5. PMID 33151090
- [Background] Kearns SM, Ahern KW, Patrie JT, Horton WB, Harris TE, Kadl A. Reduced adiponectin levels in patients with COVID-19 acute respiratory failure: A case-control study. Physiol Rep. 2021 Apr;9(7):e14843. doi: 10.14814/phy2.14843. PMID 33904656
- [Background] Fukushima A, Kinugawa S, Homma T, Masaki Y, Furihata T, Yokota T, Matsushima S, Abe T, Suga T, Takada S, Kadoguchi T, Katsuyama R, Oba K, Okita K, Tsutsui H. Decreased serum brain-derived neurotrophic factor levels are correlated with exercise intolerance in patients with heart failure. Int J Cardiol. 2013 Oct 12;168(5):e142-4. doi: 10.1016/j.ijcard.2013.08.073. Epub 2013 Aug 27. No abstract available. PMID 24029660
- [Background] Kirwan R, McCullough D, Butler T, Perez de Heredia F, Davies IG, Stewart C. Sarcopenia during COVID-19 lockdown restrictions: long-term health effects of short-term muscle loss. Geroscience. 2020 Dec;42(6):1547-1578. doi: 10.1007/s11357-020-00272-3. Epub 2020 Oct 1. PMID 33001410
- [Background] Sagarra-Romero L, Vinas-Barros A. COVID-19: Short and Long-Term Effects of Hospitalization on Muscular Weakness in the Elderly. Int J Environ Res Public Health. 2020 Nov 24;17(23):8715. doi: 10.3390/ijerph17238715. PMID 33255233
- [Background] Nobari H, Fashi M, Eskandari A, Perez-Gomez J, Suzuki K. Potential Improvement in Rehabilitation Quality of 2019 Novel Coronavirus by Isometric Training System; Is There "Muscle-Lung Cross-Talk"? Int J Environ Res Public Health. 2021 Jun 10;18(12):6304. doi: 10.3390/ijerph18126304. PMID 34200791